CLINICAL TRIAL: NCT00443612
Title: A Randomized, Open Label, Cross-over Comparative Study of Irbesartan/Hydrochlorothiazide and Irbesartan in the Treatment of Mild to Moderate Hypertension
Brief Title: Irbesartan/Hydrochlorothiazide National Taiwan University Hospital Listing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRBEH_L_00702
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan; Hydrochlorothiazide

ARMS (2):
- 1 (Experimental): * 12 weeks on treatment 1
  * 2 week washout period
  * 12 weeks on treatment 2
  Interventions: Drug: Irbesartan/Hydrochlorothiazide; Drug: Irbesartan
- 2 (Experimental): * 12 weeks on treatment 2
  * 2 week washout period
  * 12 weeks on treatment 1
  Interventions: Drug: Irbesartan/Hydrochlorothiazide; Drug: Irbesartan

INTERVENTIONS:
Drug: Irbesartan/Hydrochlorothiazide — Administration of irbesartan 150 mg/day + hydrochlorothiazide 12.5 mg
Drug: Irbesartan — Administration of irbesartan 150 mg/day

SUMMARY:
Primary:

1. To compare the change in forearm vascular resistance following a 12-week regimen of irbesartan/hydrochlorothiazide versus irbesartan
2. To assess changes of serum proinflammatory cytokine, markers of cardiovascular risks, oxidative stress and circulating adhesion molecule including thiobarbiturate acid reactive substances (TBARS), C-reactive protein (CRP), interleukin 6 (IL-6), and vascular cell adhesion molecule 1 (VCAM-1).

Secondary:

1. To compare the reduction in office blood pressure following a 12-week regimen of irbesartan/hydrochlorothiazide versus irbesartan
2. To compare the response rate (defined as office Systolic blood pressure(SBP)/diastolic blood pressure (DBP) reduce more than 10mmHg from baseline), and BP controlled rate (defined as SBP<140 mmHg and /or DBP<90 mmHg)
3. To ascertain the safety and tolerability of irbesartan / hydrochlorothiazide versus irbesartan when administered once daily
4. To determine whether angiotensin II type 1 (AT-1) receptor gene polymorphisms (including A1166C gene with about 4% of the minor allele frequency in Chinese population and other single nucleotide polymorphisms with a higher frequency of about 10% of minor allele) is related to reduction of BP

ELIGIBILITY:
Inclusion Criteria:

Patients with mild to moderate hypertension with office diastolic BP (DBP) 90-109 mmHg and/or systolic BP (SBP) 140-179 mmHg before entering each treatment

Exclusion Criteria:

* females: who are pregnant or breast feeding
* office DBP ≧ 110 mmHg or office SBP ≧ 180 mmHg
* history of significant cardiovascular diseases which include: acute myocardial infarction within six months or any ischemic heart disease requiring medication, or cerebrovascular disease
* history of significant renal diseases including: serum creatinine > 3.0 mg/dl, or creatinine clearance < 30 ml/min.
* severe biliary cirrhosis and cholestasis
* refractory hypokalemia, hypercalcemia
* history of autoimmune disease, collagen vascular disease, multiple drug allergies, bronchospastic disease or other malignancies requiring current medication
* hepatic disease as indicated by any of the following : Serum Glutamic Oxaloacetic Transaminase (SGOT) or Serum Glutamic Pyruvate Transaminase (SGPT) >3 x upper limit of normal, or serum bilirubin > 2 x upper limit of normal

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Forearm vascular resistance | At baseline and end of study
Changes of serum TBARS, CRP, IL-6, and VCAM-1 | Throughout the study period
Office BP measurement of seated SBP and DBP | At baseline and after 12-week treatment
Adverse events | Throughout the study period

SECONDARY OUTCOMES:
Office BP measurement of seated SBP and DBP | At baseline and after 12-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fern Lim, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Taipei, Taiwan